CLINICAL TRIAL: NCT00082628
Title: A Phase III, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Safety and Efficacy of Serostim®, r-hGH in the Treatment and Maintenance of Human Immunodeficiency HIV-Associated Adipose Redistribution Syndrome, or HARS
Brief Title: Treatment of Abnormal Adipose Tissue Accumulation in Human Immunodeficiency Virus (HIV) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24380
Record Dates: First submitted 2004-05-13; First posted 2004-05-17 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-09

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: Growth hormone; Serostim®; Human Adipose Redistribution Syndrome; Human Immunodeficiency Virus lipodystrophy
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Period I: Placebo (Placebo Comparator): Subjects will receive placebo matched to serostim® as subcutaneous injection daily for a period of 12 weeks.
  Interventions: Drug: Placebo
- Period I: Serostim® 4 mg (Experimental): Subjects will receive Serostim® as subcutaneous injection at a maximum dose of 4 milligram (mg) per day based on body weight for a period of 12 weeks.
  Interventions: Drug: Serostim® 4 mg
- Period II: Serostim® 4 mg to Placebo (Experimental): All subjects who will be initially randomized to Serostim® 4 mg arm in Period I and will receive placebo matched to Serostim® on alternate days for 24 weeks in Period II.
  Interventions: Drug: Placebo
- Period II: Serostim® 4 mg to Serostim® 2 mg (Experimental): All subjects who will be initially randomized to Serostim® 4 mg arm in Period I and will receive Serostim® 2 mg on alternate days for 24 weeks in Period II.
  Interventions: Drug: Serostim® 2 mg
- Period II: Placebo to Placebo/Serostim® 4 mg (Experimental): All subjects who will be initially randomized to Placebo arm in Period I continue receiving placebo matched to Serostim® on alternate days for 12 weeks followed by Serostim® 4 mg daily 12 weeks.
  Interventions: Drug: Placebo; Drug: Serostim® 4 mg

INTERVENTIONS:
Drug: Placebo — Placebo matched to serostim® as subcutaneous injection.
  Arms: Period I: Placebo; Period II: Placebo to Placebo/Serostim® 4 mg; Period II: Serostim® 4 mg to Placebo
Drug: Serostim® 4 mg — Serostim® as subcutaneous injection at a maximum dose of 4 milligram (mg) per day based on body weight.
  Other Names: recombinant human growth hormone (r-hGH)
  Arms: Period I: Serostim® 4 mg; Period II: Placebo to Placebo/Serostim® 4 mg
Drug: Serostim® 2 mg — Serostim® 2 mg as subcutaneous injection on alternate days.
  Other Names: recombinant human growth hormone (r-hGH)
  Arms: Period II: Serostim® 4 mg to Serostim® 2 mg

SUMMARY:
The primary objective of the study is to determine if Serostim® 4 mg administered daily for 12 weeks as treatment for the abnormal fat accumulation and distribution associated with HIV-associated Adipose Redistribution Syndrome (HARS) reduces Visceral Adipose Tissue (VAT, measured by CT scan) more effectively than placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Have written laboratory documentation of an HIV infection by one of the following methods:

   * Detectable viral load measured by polymerase chain reaction (PCR) amplification, branched chain DNA (bDNA) signal amplification or the presence of p24 antigen.
   * Presence of HIV antibodies confirmed by either Western blot or immunofluorescence assay.

   Written laboratory documentation of an HIV infection must be obtained prior to randomization. In the absence of documented historical confirmation, an assay of HIV antibodies will be included in the Screening Laboratory Panel. Results will be confirmed with a Western Blot.
2. Have evidence of excess abdominal adipose deposition when measured by the anthropometric methodology, using the following cut off values:

   * Men: Waist circumference >88.2 cm AND waist: hip ratio >= 0.95.
   * Women: Waist circumference >75.3 cm AND waist: hip ratio >= 0.9.
3. Are taking antiretroviral medication(s) which is (are) approved or is (are) available under a Treatment IND. The regimen must have remained stable for 30 days prior to study entry. Subjects must also agree not to discontinue or to change their regimen for the duration of the study except as judged medically necessary.
4. Have parameter values less than the following limits (using results from the central laboratory):

   * AST, ALT, and amylase <= 3 times the upper limit of normal (Screening).
   * Fasting triglycerides <= 1,000 mg/dL (Screening).
   * Fasting glucose <110 mg/dL (Screening).
   * Two-hour (120 minute) glucose <140 mg/dL (Screening).
5. Weight >= 36 kg (79.3 lb)
6. Be between 18 and 60 years of age (inclusive) unless local law dictates different limits.
7. Sufficiently literate in English to be able to comprehend and complete the Quality of Life Questionnaire.
8. Willing and able to comply with the protocol for the duration of the study.
9. Have voluntarily provided written informed consent (with subject authorization under HIPAA), prior to performing any study-related procedure that is not part of normal medical care, and with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
10. Female subjects must:

    1. Be post menopausal (>= 1 year) or surgically sterilized (i.e., have undergone tubal ligation or hysterectomy)

       or
    2. Use a contraceptive method for the duration of the study such as:

       * Hormonal contraceptive
       * Intra uterine device
       * Diaphragm with spermicide, or condom with spermicide.

       And
    3. Must be neither pregnant nor breast feeding.
    4. Confirmation that female subjects of childbearing potential are not pregnant must be established by a negative beta-hCG serum pregnancy test during the 14-day screening period prior to Study Day 1. If the beta-hCG serum pregnancy test is performed more than 7 days prior to Study Day 1, a urine pregnancy test must be performed by the site laboratory on Study Day 1 to confirm a negative test result.

Exclusion Criteria:

1. Have an active AIDS-defining opportunistic complication (OC) as defined by the CDC or have had an untreated or suspected serious systemic infection, or have had a persistent fever >= 101°F (38.3°C) during the 30 days prior to study entry.
2. Any active or past history of malignancy, except for localized cutaneous Kaposi's sarcoma (fewer than 10 lesions, none of which are larger than 2 cm, and not on active therapy). Such exceptions must be confirmed in writing by the Serono Study Director.
3. Have a CNS mass or active CNS process associated with neurological findings.
4. Have unstable or untreated hypertension, defined as >= 140/90 mm Hg at the time of the Screening Visit, and/or have initiated or changed antihypertensive therapy in the 30 days prior to Study Day 1.
5. Have an acute critical illness treated in an intensive care unit, e.g., due to complications following open heart or abdominal surgery, multiple accidental trauma, or acute respiratory failure.
6. Have a recent history of sleep apnea or intermittent upper respiratory obstruction.
7. Have any condition, which interferes with informed consent or protocol compliance including, but not limited to, active substance abuse and/or dementia.
8. Are unable to comply with the Concomitant Therapy restrictions including:

   * therapy for obesity including therapy with anorexigenic or fat reducing drugs
   * anti-diabetic or insulin sensitizing medications
   * systemic glucocorticoids
   * systemic chemotherapy, interferon or radiation therapy treatment
   * androgenic agents including, but not limited to testosterone, nandrolone, oxandrolone, oxymetholone, etc. (testosterone replacement therapy for hypogonadism is the exception to this exclusion and will be allowed if started > 30 days prior to Study Day 1)
   * progestational agents, unless used for oral contraception or post-menopausal hormone replacement therapy
   * appetite stimulants
   * investigational agents, unless approved in advance by the study medical director. Specifically, experimental antiretroviral agents are disallowed, unless available under a treatment IND or expanded access program (30 days).
   * Liposuction or other elective plastic surgery
   * AIDS wasting therapy or prior growth hormone treatment other than study drug (for 12 months prior to the screening visit)
9. Have ever been diagnosed with any of the following conditions:

   * Pancreatitis
   * Carpal tunnel syndrome (unless resolved by surgical release)
   * Diabetes mellitus
   * Angina pectoris
   * Coronary artery disease
   * Any disorder associated with moderate to severe edema (e.g., ascites, nephrotic syndrome, congestive heart failure, lymphedema).
10. Allergy or hypersensitivity to growth hormone.
11. Are participating in any other clinical studies.

In order to participate in this trial a subject must meet all of the inclusion and exclusion criteria specified above. Requests for protocol exceptions/exemptions must come from a participating, fully initiated site at which a prospective patient has consented to undergo screening. Exceptions/exemptions are only allowed by the Trial Director. There is no program in place to allow drug for a single patient IND, or for an expanded access protocol. This statement holds true for both children and adults.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2004-05-28 (Actual); Primary Completion 2005-09-28 (Actual); Study Completion 2005-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (31):
- United States (30):
  - University of Alabama/Birmingham, Birmingham, Alabama
  - CARE CLINIC - UCLA Medical Center, Los Angeles, California
  - 1401 N. Palm Canyon, Palm Springs, California
  - Trials Unit Div of Infectious and Immunologic Diseases, Sacramento, California
  - UCSD - AntiViral Research Center, San Diego, California
  - University of California, San Francisco - Div. of Endocrinology, San Francisco, California
  - Kaiser Permanente, San Francisco, California
  - Northern California Institute for Research and Education, Inc., San Francisco, California
  - Harbor-UCLA Medical Ctr Research & Education Institute, Torrance, California
  - AIDS Alliance, West Hollywood, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - 1640 Rhode Island Avenue, N.W., Washington D.C., District of Columbia
  - Office Of Dr Gary Richmond, Fort Lauderdale, Florida
  - 3661 South Miami Avenue, Miami, Florida
  - Care Resources, Miami, Florida
  - Infectious Disease Associates, Sarasota, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tufts University School of Medicine, Boston, Massachusetts
  - Community Research Initiative of New England, Boston, Massachusetts
  - Community Research Initiative Of New England, Springfield, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Albany Medical College, Albany, New York
  - Weill Medical College of Cornell Universtiy, New York, New York
  - St. Luke's Roosevelt Hospital, New York, New York
  - Bronx Women's Interagency HIV Study, The Bronx, New York
  - Central Texas Clincial research, Austin, Texas
  - IDP Research, Annandale, Virginia
  - Office of Daniel Coulston, M.D., Spokane, Washington
- AIDS Research Program, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.serostim.com
- See also: Link to PubMed — http://www.ncbi.nlm.nih.gov/pubmed/17592343?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=1
- See also: Related Info — http://journals.lww.com/jaids/Fulltext/2007/07010/Recombinant_Human_Growth_Hormone_to_Treat.6.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Period I: Placebo: Subjects received placebo matched to serostim® as subcutaneous injection daily for a period of 12 weeks.
- Period I: Serostim® 4 mg: Subjects received Serostim® as subcutaneous injection at a maximum dose of 4 milligram (mg) per day based on body weight for a period of 12 weeks.
- Period II: Serostim® 4 mg to Placebo: All subjects who were initially randomized to Serostim® 4 mg arm in Period I and received placebo matched to Serostim® on alternate days for 24 weeks in Period II.
- Period II: Serostim® 4 mg to Serostim® 2 mg: All subjects who were initially randomized to Serostim® 4 mg arm in Period I and received Serostim® 2 mg on alternate days for 24 weeks in Period II.
- Period II: Placebo to Placebo/Serostim® 4 mg: All subjects who were initially randomized to Placebo arm in Period I continued receiving placebo matched to Serostim® on alternate days for 12 weeks followed by Serostim® 4 mg daily 12 weeks.
Period: Treatment Period I (Week 1 to Week 12)
Arm/Group | Period I: Placebo | Period I: Serostim® 4 mg | Period II: Serostim® 4 mg to Placebo | Period II: Serostim® 4 mg to Serostim® 2 mg | Period II: Placebo to Placebo/Serostim® 4 mg
Started | 81 | 245 | 0 | 0 | 0
Completed | 73 | 185 | 0 | 0 | 0
Not Completed | 8 | 60 | 0 | 0 | 0
Not completed — Subjects Did Not Receive Study Drug | 0 | 1 | 0 | 0 | 0
Not completed — Subjects Without Post-Baseline Assessmen | 2 | 1 | 0 | 0 | 0
Not completed — Subjects Did Not Complete Week 12 | 5 | 43 | 0 | 0 | 0
Not completed — Did not continue to Period II | 1 | 15 | 0 | 0 | 0
Period: Treatment Period II: Week 12 to Week 36
Arm/Group | Period I: Placebo | Period I: Serostim® 4 mg | Period II: Serostim® 4 mg to Placebo | Period II: Serostim® 4 mg to Serostim® 2 mg | Period II: Placebo to Placebo/Serostim® 4 mg
Started | 0 | 0 | 93 | 92 | 73
Completed | 0 | 0 | 78 | 76 | 55
Not Completed | 0 | 0 | 15 | 16 | 18
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Subjects Did Not Complete Week 36 | 0 | 0 | 15 | 15 | 17

BASELINE CHARACTERISTICS:
Population: The modified ITT Population (ITT) for Period I was defined as all subjects who had a baseline and at least one post-baseline efficacy measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Period I: Placebo | Period I: Serostim® 4 mg | Total
Number analyzed (Participants) | 79 | 243 | 322
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (7.5) | 44.5 (7.0) | 44.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 36 | 47
  Male | 68 | 207 | 275

OUTCOME MEASURES:

1. Primary Outcome: Treatment Period I: Change From Baseline in Absolute Area of Visceral Adipose Tissue (VAT) at Week 12
Description: Absolute area of VAT was measured by cross-sectional computed tomography (CT) scan at the level of the L4-5 inter-vertebral disk. CT scanning was to be used to assess the cross sectional area of abdominal fat and its distribution between the visceral and subcutaneous compartments, as measured at L4-L5.
Time Frame: Baseline, Week 12
Population: The modified ITT Population was defined as all subjects who had a baseline and at least one post-baseline efficacy measurement in treatment period I. Here "Overall Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Square Centimeter (cm^2)
Arm/Group | Period I: Placebo | Period I: Serostim® 4 mg
Number analyzed (Participants) | 74 | 210
Square Centimeter (cm^2) | 0.5 (34.5) | -32.6 (37.9)
Statistical Analysis 1: Comparison: Period I: Placebo vs Period I: Serostim® 4 mg; Test type: Superiority or Other; p < 0.001, Nonparametric ANCOVA Model

2. Secondary Outcome: Treatment Period I: Change From Baseline in Trunk Fat at Week 12
Description: Changes in trunk fat was measured as changes in mass (kg) on Dual-Energy X-Ray Absorptiometry (DXA) Scan.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Period I: Placebo | Period I: Serostim® 4 mg
Number analyzed (Participants) | 75 | 213
Kilogram (Kg) | 0.2 (1.3) | -2.2 (1.7)

3. Secondary Outcome: Change From Baseline in Patient Reported Outcome of Body Image Distress at Week 12
Description: Body image distress was assessed on a scale ranging from 0 to 100, where 0 = Extremely Upsetting and 100 = Extremely Encouraging.
Time Frame: Baseline, Week 12
Population: The modified ITT Population was defined as all subjects who had a baseline and at least one post-baseline efficacy measurement in treatment period I.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period I: Placebo | Period I: Serostim® 4 mg
Number analyzed (Participants) | 79 | 243
units on a scale | 0.23 (1.42) | 0.10 (1.73)

4. Secondary Outcome: Treatment Period I: Change From Baseline in Non- High-density Lipoprotein (Non-HDL) Cholesterol at Week 12
Description: Lipid profile data was analyzed for Non-HDL Cholesterol.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Period I: Placebo | Period I: Serostim® 4 mg
Number analyzed (Participants) | 74 | 226
milligram/deciliter (mg/dL) | -2.8 (28.1) | -13.0 (37.1)

5. Secondary Outcome: Treatment Period II: Failure Rate at Week 36 Based on Visceral Adipose Tissue (VAT) For Subjects Who Received Serostim® 4 mg in Period I
Description: Failure rate based on VAT was assessed by CT scan at L4-L5. The failure rate was defined as the percentage of subjects who regained >50% of their VAT lost in Treatment Period I. This outcome was to be assessed for subjects who received Serostim® 4 mg in Period I.
Time Frame: Week 36
Population: The modified ITT Population for treatment period II was defined as subjects who were re-randomized into Weeks 12 to 36 of the study and who had at least one post-Week 12 efficacy evaluation. Here "Overall Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | Period II: Serostim® 4 mg to Placebo | Period II: Serostim® 4 mg to Serostim® 2 mg
Number analyzed (Participants) | 83 | 75
percentage of subjects | 53.7 | 40.3

ADVERSE EVENTS:
Description: Safety analyses were performed on subjects who received at least one injection of study drug (Serostim® or placebo).
Groups:
- Period I: Placebo (Week 1 to 12): Subjects received placebo matched to serostim® as subcutaneous injection daily for a period of 12 weeks.
- Period I: Serostim® 4 mg (Week 1 to 12): Subjects received serostim® as subcutaneous injection at a maximum dose of 4 milligram (mg) per day based on body weight for a period of 12 weeks.
- Period II: Serostim® 4 mg to Placebo (Week 12 to 36): All subjects who were initially randomized to Serostim® 4 mg arm in Period I and received placebo matched to Serostim® on alternate days for 24 weeks in Period II.
- Period II: Serostim® 4 mg to Serostim® 2 mg (Week 12 to 36): All subjects who were initially randomized to Serostim® 4 mg arm in Period I and received Serostim® 2 mg on alternate days for 24 weeks in Period II.
- Period II: Placebo to Placebo (Week 12 to Week 24): All subjects who were initially randomized to Placebo arm in Period I continued receiving placebo matched to Serostim® on alternate days for 12 weeks in Period II.
- Period II: Placebo to Serostim® 4 mg (Week 24 to 36): All subjects who were initially randomized to Placebo arm in Period I and received Serostim® 4 mg daily 12 weeks in Period II.
Arm/Group | Period I: Placebo (Week 1 to 12) | Period I: Serostim® 4 mg (Week 1 to 12) | Period II: Serostim® 4 mg to Placebo (Week 12 to 36) | Period II: Serostim® 4 mg to Serostim® 2 mg (Week 12 to 36) | Period II: Placebo to Placebo (Week 12 to Week 24) | Period II: Placebo to Serostim® 4 mg (Week 24 to 36)
Serious Adverse Events (participants affected / at risk) | 2/81 | 3/244 | 3/93 | 2/92 | 2/73 | 1/73
Other Adverse Events (participants affected / at risk) | 70/81 | 244/244 | 46/93 | 48/92 | 14/73 | 73/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period I: Placebo (Week 1 to 12) (N=81) | Period I: Serostim® 4 mg (Week 1 to 12) (N=244) | Period II: Serostim® 4 mg to Placebo (Week 12 to 36) (N=93) | Period II: Serostim® 4 mg to Serostim® 2 mg (Week 12 to 36) (N=92) | Period II: Placebo to Placebo (Week 12 to Week 24) (N=73) | Period II: Placebo to Serostim® 4 mg (Week 24 to 36) (N=73)
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic insufficiency (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period I: Placebo (Week 1 to 12) (N=81) | Period I: Serostim® 4 mg (Week 1 to 12) (N=244) | Period II: Serostim® 4 mg to Placebo (Week 12 to 36) (N=93) | Period II: Serostim® 4 mg to Serostim® 2 mg (Week 12 to 36) (N=92) | Period II: Placebo to Placebo (Week 12 to Week 24) (N=73) | Period II: Placebo to Serostim® 4 mg (Week 24 to 36) (N=73)
Oedema peripheral (General disorders) | 4 | 113 | 4 | 6 | 0 | 34
Arthralgia (General disorders) | 14 | 95 | 5 | 8 | 2 | 30
Pain in extremity (General disorders) | 3 | 46 | 5 | 2 | 2 | 19
Headache (General disorders) | 3 | 39 | 4 | 5 | 0 | 8
Myalgia (General disorders) | 3 | 34 | 0 | 0 | 0 | 14
Blood glucose increased (General disorders) | 2 | 33 | 3 | 6 | 2 | 11
Hypoaesthesia (General disorders) | 0 | 34 | 1 | 5 | 0 | 8
Paraesthesia (General disorders) | 3 | 25 | 0 | 0 | 1 | 5
Fatigue (General disorders) | 1 | 23 | 0 | 0 | 0 | 6
Insomnia (General disorders) | 2 | 22 | 0 | 0 | 0 | 0
Joint stiffness (General disorders) | 0 | 22 | 0 | 0 | 1 | 4
Back pain (General disorders) | 4 | 15 | 0 | 0 | 1 | 3
Musculoskeletal stiffness (General disorders) | 1 | 18 | 0 | 0 | 1 | 9
Upper respiratory tract infection (General disorders) | 6 | 13 | 15 | 7 | 0 | 0
Hyperglycaemia (General disorders) | 1 | 17 | 0 | 0 | 2 | 10
Nausea (General disorders) | 3 | 15 | 0 | 0 | 1 | 3
Joint swelling (General disorders) | 0 | 17 | 0 | 0 | 0 | 5
Fluid retention (General disorders) | 0 | 13 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 6 | 7 | 0 | 0 | 0 | 0
Diarrhoea (General disorders) | 5 | 7 | 8 | 4 | 0 | 0
Nasopharyngitis (General disorders) | 5 | 6 | 1 | 5 | 0 | 0
Sinusitis (General disorders) | 4 | 6 | 0 | 0 | 0 | 0
Muscle spasms (General disorders) | 0 | 0 | 0 | 0 | 0 | 4
Shoulder pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 4
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other